CLINICAL TRIAL: NCT03502733
Title: Phase Ib Study of Copanlisib in Combination With Nivolumab or With Nivolumab and Ipilimumab
Brief Title: Testing the Combination of Copanlisib, Nivolumab and Ipilimumab in Patients With Advanced Cancer and Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-02249; NCI-2017-02249 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI CC 18-C-0122; 10145 (Other: National Cancer Institute LAO); 10145 (Other: CTEP); ZIABC011078 (NIH)
Record Dates: First submitted 2018-04-17; First posted 2018-04-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma; Metastatic Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Lymphoma; Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; copanlisib; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort I (Doublet) (copanlisib, nivolumab) (Experimental): Patients receive copanlisib IV over 1 hour on days 1 and 15 or days 1, 8, and 15 of each cycle and nivolumab IV over 30 minutes on day 1 or days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan and/or MRI throughout the trial. Patients undergo blood sample collection on study and during follow-up, as well as tumor biopsy on study. Patients also undergo an ECHO during screening and as clinically indicated on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Copanlisib; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab
- Cohort II (Triplet Safety) (copanlisib, nivolumab, ipilimumab) (Experimental): Patients receive copanlisib IV over 1 hour on days 1, 8, and 15 of each cycle, nivolumab IV over 30 minutes on day 1 of each cycle, and ipilimumab IV over 90 minutes on day 1 for cycles 1-4. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan and/or MRI throughout the trial. Patients undergo an ECHO during screening and as clinically indicated on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Copanlisib; Procedure: Echocardiography Test; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab
- Cohort III (Triplet) (copanlisib, nivolumab, ipilmumab) (Experimental): Patients receive copanlisib IV over 1 hour on days 1, 8, and 15 of each cycle, nivolumab IV over 30 minutes on day 15 of cycle 1 and then day 1 of each subsequent cycles, and ipilimumab IV over 90 minutes on day 1 for cycles 2-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan and/or MRI throughout the trial. Patients undergo blood sample collection on study and during follow-up, as well as tumor biopsy on study. Patients also undergo an ECHO during screening and as clinically indicated on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Copanlisib; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Copanlisib — Given IV
  Other Names: BAY 80 6946; BAY 80-6946; BAY 806946; BAY-80-6946; BAY806946; PI3K Inhibitor BAY 80-6946
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Cohort II (Triplet Safety) (copanlisib, nivolumab, ipilimumab)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase Ib trial studies the side effects and best dose of copanlisib and nivolumab and side effects of copanlisib given together with nivolumab and ipilimumab in treating patients with solid tumors that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or lymphoma. Copanlisib stops tumors from growing by blocking proteins that are known to be important for tumor cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving copanlisib together with nivolumab or with nivolumab and ipilimumab may work better in treating patients with solid tumors or lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the safety, tolerability, and the recommended phase 2 dose (RP2D) of copanlisib and nivolumab combination in patients with advanced solid tumors and lymphomas.

II. To evaluate the safety and tolerability of copanlisib combined with nivolumab and ipilimumab in patients with advanced solid tumors and lymphomas.

EXPLORATORY OBJECTIVES:

I. Evaluate the effect of the doublet and triplet combinations on markers of anti-tumor immunity in circulating immune cells and pre- and post-treatment tumor biopsies.

II. Evaluate the effect of the combinations on biomarkers of AKT inhibition, deoxyribonucleic acid (DNA) damage (gammaH2AX, pNbs1, Rad51), apoptosis, and epithelial-mesenchymal transition in pre- and post- treatment tumor biopsies.

III. Assess preliminary antitumor activity of the combinations.

OUTLINE: This is a dose-escalation study of copanlisib and nivolumab, followed by a dose-expansion study.

COHORT I (DOUBLET TREATMENT PLAN): Patients receive copanlisib intravenously (IV) over 1 hour on days 1 and 15 or days 1, 8, and 15 of each cycle and nivolumab IV over 30 minutes on day 1 or days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) scan and/or magnetic resonance imaging (MRI) throughout the trial. Patients undergo blood sample collection on study and during follow-up, as well as tumor biopsy on study. Patients also undergo an echocardiography (ECHO) during screening and as clinically indicated on study.

COHORT II (TRIPLET SAFETY RUN-IN PHASE TREATMENT PLAN): Patients receive copanlisib IV over 1 hour on days 1, 8, and 15 of each cycle, nivolumab IV over 30 minutes on day 1 of each cycle, and ipilimumab IV over 90 minutes on day 1 for cycles 1-4. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan and/or MRI throughout the trial. Patients undergo an ECHO during screening and as clinically indicated on study.

COHORT III (TRIPLET TREATMENT PLAN): Patients receive copanlisib IV over 1 hour on days 1, 8, and 15 of each cycle, nivolumab IV over 30 minutes on day 15 of cycle 1 and then day 1 of each subsequent cycles, and ipilimumab IV over 90 minutes on day 1 for cycles 2-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan and/or MRI throughout the trial. Patients undergo blood sample collection on study and during follow-up, as well as tumor biopsy on study. Patients also undergo an ECHO during screening and as clinically indicated on study.

After completion of study treatment, patients are followed up monthly for 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented metastatic, recurrent, or locally unresectable solid tumors which have progressed after one line of therapy, or for which no curative therapy is available. Patients with lymphoma who have received adequate exposure to standard of care therapy and for whom no curative therapy is available are also eligible (this trial will enroll a minimum of 5 lymphoma patients)
* Patients must have measurable or evaluable disease
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Leukocytes >= 2,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL (solid tumor patients) >= 75,000/mcL (lymphoma patients)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) /alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional ULN
* Serum creatinine =< 1.5 x institutional ULN OR creatinine clearance >= 50 mL/min/1.73 m^2 by Cockcroft-Gault
* Any prior therapy must have been completed >= 4 weeks (6 weeks for nitrosoureas and mitomycin C) or, if known, >= 5 half-lives of the prior agent (whichever is shorter) prior to enrollment on protocol (minimum of 1 week between prior therapy and study enrollment), and the participant must have recovered to eligibility levels from prior toxicity; prior definitive radiation should have been completed >= 4 weeks or palliative radiation should have been completed >= 2 weeks prior to study enrollment and all associated toxicities resolved to eligibility levels (patients on study may be eligible for palliative radiotherapy to non-targeted lesions after 2 cycles of therapy at the principal investigator's [PI's] discretion); patients must be >= 2 weeks since any investigational agent administered as part of a phase 0 study (where a sub-therapeutic dose of drug is administered) at the PI's discretion, and should have recovered to grade 1 or baseline from any toxicities
* Patients who have had prior monoclonal antibody therapy must have completed that therapy >= 6 weeks (or 3 half-lives of the antibody, whichever is shorter) prior to enrollment on protocol (minimum of 1 week between prior therapy and study enrollment)
* Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that their medication dose is stable, and international normalized ratio/partial thromboplastin time (INR/PTT) remains stable within the recommended therapeutic range
* Patients must have left ventricular ejection fraction (LVEF) >= 50%
* The effects of nivolumab, copanlisib and ipilimumab on the developing human fetus are unknown, and there is potential for teratogenic or abortifacient effects. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the treatment portion of the study, and for a minimum of 5 months after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to study entry, for the duration of study participation, and for 7 months after completion of study treatment
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to provide blood for research purposes (all patients, apart from patients enrolled onto triplet safety run-in phase) and willingness to provide new tumor biopsy samples for research purposes (doublet and triplet expansion cohorts)

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* Patients with clinically significant illnesses which would compromise participation in the study, including but not limited to active or uncontrolled infection, immune deficiencies, hepatitis B, hepatitis C, active tuberculosis, uncontrolled asthma, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, myocardial infarction within the past 6 months, cerebral vascular accident/stroke within the past 6 months, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with known brain metastases or carcinomatous meningitis are excluded from this clinical trial, with the exception of patients whose brain metastatic disease status has remained stable for >= 1 month after treatment of the brain metastases; patients on anti-seizure medications may be enrolled at the discretion of the principal investigator
* Patients with blood oxygen saturation < 90% at rest; patients must not have symptomatic interstitial lung disease, pneumonitis, or known pulmonary fibrosis. Patients must also not have a history of interstitial lung disease of any severity
* Patients with uncontrolled arterial hypertension are ineligible. Uncontrolled arterial hypertension is defined as an average blood pressure of > 140 mm Hg systolic and/or > 90 mm Hg diastolic over 3 measurements, taken over the course of one clinic visit at intervals of >=30 minutes. Patients with well-controlled arterial hypertension are eligible
* Patients with uncontrolled Type I or II diabetes mellitus, defined as fasting blood glucose of > 160 mg/dL and glycosylated hemoglobin measurement (HgA1c) > 8.5%, are ineligible. Patients with fasting blood glucose >160 mg/dL may be eligible if the HgA1c < 8.5%, per PI discretion. Patients with well-controlled diabetes mellitus are eligible
* Patients are not eligible if they have had or are planned for solid organ transplant or allogeneic hematopoietic stem cell transplant
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; however, systemic corticosteroids may be indicated after starting the study drugs to treat immune-related adverse reactions; inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Doublet cohort and triplet safety run-in phase: Patients are not eligible if they have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting immune checkpoint pathways. Patients should therefore be excluded if they have had prior treatment with the combination of a PI3K inhibitor and a PD-1 inhibitor; however, prior treatment with a PI3K/AKT/mTOR inhibitor (without the addition of a checkpoint inhibitor) is allowed. Patients that have had prior chimeric antigen receptor (CAR) T-cell therapy are eligible
* Triplet pharmacodynamic phase only: Patients who have previously received one line of immunotherapy (including checkpoint inhibitors) are eligible; however, patients previously receiving ipilimumab + nivolumab combination therapy are excluded. Patients who received prior therapy with a checkpoint inhibitor and were taken off drug for serious adverse events are excluded. Prior treatment with a PI3K/AKT/mTOR inhibitor, or prior CAR T-cell therapy is allowed
* Copanlisib is primarily metabolized by CYP3A4. Therefore, the concomitant use of strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir) and strong inducers of CYP3A4 (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, St. John's Wort) is not permitted from 14 days prior to enrollment until the end of the study. Other medications that are prohibited while on copanlisib treatment:

  * Herbal medications/preparations (except for vitamins)
  * Anti-arrhythmic therapy other than beta blockers or digoxin
* Human immunodeficiency virus (HIV)-positive patients are eligible if on stable dose of highly active antiretroviral therapy (HAART), no clinically significant drug-drug interactions are anticipated with the current HAART regimen, and viral load is undetectable. Patients on HAART regimens that include CYP3A4 inhibitors (e.g. ritonavir or cobicistat) are excluded. All patients must be screened for HIV up to 28 days prior to enrollment
* Hepatitis B (HBV) or hepatitis C (HCV) infection. All patients must be screened for HBV and HCV up to 28 days prior to enrollment using the routine hepatitis virus lab panel. Patients positive for hepatitis B virus surface antigen measurement (HBsAg) and/or hepatitis B virus core antibody measurement (HBcAb) will be eligible if they are negative for HBV DNA; these patients should receive prophylactic antiviral therapy. Patients positive for anti-HCV antibody will be eligible if they are negative for HCV ribonucleic acid (RNA)
* Cytomegalovirus (CMV) infection. All patients must be screened for CMV up to 28 days prior to enrollment. Patients that are positive for CMV DNA by polymerase chain reaction (PCR) are not eligible for the study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to copanlisib, PI3K inhibitors, nivolumab, or ipilimumab
* Patients with active autoimmune disease requiring systemic treatment within the past 3 months, a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents are not eligible. Patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Patients that require intermittent use of bronchodilators or local steroid injections will not be excluded from the study. Patients with hypothyroidism and stable on hormone replacement or Sjogren's syndrome will not be excluded from the study
* Pregnant or breastfeeding women will be excluded from participation in this trial, as there is no significant preclinical information regarding the effects of nivolumab, copanlisib, and ipilimumab, on a fetus or newborn infant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-08-14 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose of copanlisib and nivolumab combination | Up to 28 days
  Will be defined as dose limiting toxicity in =< 1 out of 6 patients at highest dose level below the maximally administered dose.
Incidence of adverse events | Up to 30 days after the last dose of study drug
  Graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.

OTHER OUTCOMES:
Markers of anti-tumor immunity assessed in circulating immune cells, circulating tumor cells, and pre- and post-treatment tumor biopsies | Up to 6 years
  Evaluations will be performed, with results reported with appropriate caveats about the exploratory nature of the analysis, and without formal adjustment for multiple comparisons.
Biomarkers of AKT inhibition, deoxyribonucleic acid damage (gammaH2AX, pNbs1, Rad51), apoptosis, and epithelial-mesenchymal transition assessed in pre- and post- treatment tumor biopsies | Up to 6 years
  Evaluations will be performed, with results reported with appropriate caveats about the exploratory nature of the analysis, and without formal adjustment for multiple comparisons.
Preliminary antitumor activity | Up to 6 years
  Evaluations will be performed, with results reported with appropriate caveats about the exploratory nature of the analysis, and without formal adjustment for multiple comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: A P Chen, Principal Investigator — National Cancer Institute LAO
Locations (3):
- United States (3):
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - M D Anderson Cancer Center, Houston, Texas